CLINICAL TRIAL: NCT01860079
Title: Early Discharge After Primary Percutaneous Coronary Intervention: A Prospective Randomized Multi-center Trial (the EDAP PCI Trial)
Brief Title: Early Discharge After Primary Percutaneous Coronary Intervention
Acronym: EDAPPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: the EDAP PCI trial
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Early discharge; STEMI; PPCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early discharge group (Active Comparator): In the early discharge group, patients are actively targeted for hospital discharge within 48-56 hours.
  Interventions: Procedure: early discharge
- Standard discharge group (No Intervention): Patients who stay longer (96-120 hours) as of a standard procedure

INTERVENTIONS:
Procedure: early discharge — In the early discharge group, patients are actively targeted for hospital discharge within 48-56 hours.
  Arms: Early discharge group

SUMMARY:
* When Primary percutaneous coronary intervention (PPCI) is performed expeditiously and at a high-volume centre, it is the optimal approach for ST elevation myocardial infarction (STEMI) . In contrast to the clarity of how to treat STEMI, there is no clear definition for when to discharge and which patient to discharge.
* An early discharge strategy may be desired by all parties (financial health care provider, treating physician, nurse, patient, patient's relatives)involved in STEMI.
* The main goal in our study is to test the hypothesis that an early discharge strategy within 48-56 hours in patients with successful PPCI is as safe as in those patients who stay longer (96-120 hours) as of a standard procedure.

DETAILED DESCRIPTION:
* Primary percutaneous coronary intervention (PPCI) has become the optimal reperfusion strategy for ST elevation myocardial infarction (STEMI) when the procedure is performed expeditiously and at a high-volume centre.In contrast to the clarity of how to treat STEMI, there is no clear definition for when to discharge and which patient to discharge.
* It is conceivable to discharge patients with successful PPCI as early as possible, because a hospital stay longer than needed may create undesirable outcomes in terms of hospital infections, psychosocial reasons, adequate mobilization and patient comfort. In many tertiary centres with a busy PPCI programme insufficient bed capacity is an ongoing concern and threatens the continuous acceptance of new cases of acute infarctions. In addition, it has been indicated that an early discharge policy may lead to a substantial cost saving.
* Although much work has been done in developing and validating risk scores that identify low risk patients, data on the implementation of early discharge strategies have been quite limited There are 3 randomised trials investigating the possibility of early discharge after PPCI. However, certain limitations of these studies are preventing to implement an early discharge strategy in all-comers, particularly because of the underrepresentation of older patients in clinical trials. The verification of this policy is also needed in patients with multivessel disease. The first prospective randomized trial, the PAMI II,7 is partly obsolete as major changes have been made in PPCI with respect to devices and adjunctive medication. The other two randomized trials were single-center pilot studies with small number of patients.
* Therefore, the above mentioned literature information warrants to test the reproducibility of safety endpoints in a large scale multicenter trial, prior to application of the early discharge strategy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and subsequent written agreement of a family member (confirming good social background)
* Acute STEMI, defined as >30 minutes of continuous typical chest pain and ST-segment elevation ≥2 mm in two contiguous electrocardiography leads and /or left bundle branch block within 12 hours of symptom onset.
* Haemodynamically stable Angiographically
* Successful PPCI procedure (TIMI 2-3 flow and %<20 residual stenosis) and an uneventful 24 hour follow up period
* Single epicardial artery to be treated
* Telephone contact between the patient and PCI center after discharge is available 24 hours daily

Exclusion Criteria:

* Inability to consent
* Patients treated with thrombolytic agents for the index STEMI
* Cardiogenic shock,
* Stroke within a month,
* Signs of heart failure (Killip II-IV)
* Hypotension (<100 mmHg SBP) persisting after PPCI
* Chest pain recurrence
* Clinically significant arrhythmia (requiring treatment) occurring >6 hours after PPCI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sevket Gorgulu, MD, Study Chair — Acıbadem University School of Medicine; Tugrul Norgaz, MD, Principal Investigator — Acıbadem University School of Medicine; Sinan Dagdelen, MD, Principal Investigator — Acıbadem University School of Medicine; Nevzat Uslu, MD, Principal Investigator — Mehmet Akif Ersoy Education and Training Hospital; Aydin Yildirim, MD, Principal Investigator — Siyami Ersek Educational and Training Hospital; Ali Buturak, MD,, Principal Investigator — Acıbadem University School of Medicine
Locations (3):
- Turkey (Türkiye) (3):
  - Acibadem University, Istanbul
  - Mehmet Akif Ersoy Education and Training Hospital, Istanbul
  - Siyami Ersek Education and Training Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zijlstra F, Hoorntje JC, de Boer MJ, Reiffers S, Miedema K, Ottervanger JP, van 't Hof AW, Suryapranata H. Long-term benefit of primary angioplasty as compared with thrombolytic therapy for acute myocardial infarction. N Engl J Med. 1999 Nov 4;341(19):1413-9. doi: 10.1056/NEJM199911043411901. PMID 10547403
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Boersma E; Primary Coronary Angioplasty vs. Thrombolysis Group. Does time matter? A pooled analysis of randomized clinical trials comparing primary percutaneous coronary intervention and in-hospital fibrinolysis in acute myocardial infarction patients. Eur Heart J. 2006 Apr;27(7):779-88. doi: 10.1093/eurheartj/ehi810. Epub 2006 Mar 2. PMID 16513663
- [Background] Laarman GJ, Dirksen MT. Early discharge after primary percutaneous coronary intervention. Heart. 2010 Apr;96(8):584-7. doi: 10.1136/hrt.2009.171363. Epub 2009 Sep 23. PMID 19778921
- [Background] Newby LK, Eisenstein EL, Califf RM, Thompson TD, Nelson CL, Peterson ED, Armstrong PW, Van de Werf F, White HD, Topol EJ, Mark DB. Cost effectiveness of early discharge after uncomplicated acute myocardial infarction. N Engl J Med. 2000 Mar 16;342(11):749-55. doi: 10.1056/NEJM200003163421101. PMID 10717009
- [Background] Topol EJ, Burek K, O'Neill WW, Kewman DG, Kander NH, Shea MJ, Schork MA, Kirscht J, Juni JE, Pitt B. A randomized controlled trial of hospital discharge three days after myocardial infarction in the era of reperfusion. N Engl J Med. 1988 Apr 28;318(17):1083-8. doi: 10.1056/NEJM198804283181702. PMID 3281014
- [Background] Grines CL, Marsalese DL, Brodie B, Griffin J, Donohue B, Costantini CR, Balestrini C, Stone G, Wharton T, Esente P, Spain M, Moses J, Nobuyoshi M, Ayres M, Jones D, Mason D, Sachs D, Grines LL, O'Neill W. Safety and cost-effectiveness of early discharge after primary angioplasty in low risk patients with acute myocardial infarction. PAMI-II Investigators. Primary Angioplasty in Myocardial Infarction. J Am Coll Cardiol. 1998 Apr;31(5):967-72. doi: 10.1016/s0735-1097(98)00031-x. PMID 9561995
- [Background] Jirmar R, Widimsky P, Capek J, Hlinomaz O, Groch L. Next day discharge after successful primary angioplasty for acute ST elevation myocardial infarction. An open randomized study "Prague-5". Int Heart J. 2008 Nov;49(6):653-9. doi: 10.1536/ihj.49.653. PMID 19075481
- [Background] Kotowycz MA, Cosman TL, Tartaglia C, Afzal R, Syal RP, Natarajan MK. Safety and feasibility of early hospital discharge in ST-segment elevation myocardial infarction--a prospective and randomized trial in low-risk primary percutaneous coronary intervention patients (the Safe-Depart Trial). Am Heart J. 2010 Jan;159(1):117.e1-6. doi: 10.1016/j.ahj.2009.10.024. PMID 20102876
- [Background] Lee PY, Alexander KP, Hammill BG, Pasquali SK, Peterson ED. Representation of elderly persons and women in published randomized trials of acute coronary syndromes. JAMA. 2001 Aug 8;286(6):708-13. doi: 10.1001/jama.286.6.708. PMID 11495621
- [Background] Chesebro JH, Knatterud G, Roberts R, Borer J, Cohen LS, Dalen J, Dodge HT, Francis CK, Hillis D, Ludbrook P, et al. Thrombolysis in Myocardial Infarction (TIMI) Trial, Phase I: A comparison between intravenous tissue plasminogen activator and intravenous streptokinase. Clinical findings through hospital discharge. Circulation. 1987 Jul;76(1):142-54. doi: 10.1161/01.cir.76.1.142. PMID 3109764
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX, Anderson JL, Jacobs AK, Halperin JL, Albert NM, Brindis RG, Creager MA, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Kushner FG, Ohman EM, Stevenson WG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):e362-425. doi: 10.1161/CIR.0b013e3182742cf6. Epub 2012 Dec 17. No abstract available. PMID 23247304
- [Background] Killip T 3rd, Kimball JT. Treatment of myocardial infarction in a coronary care unit. A two year experience with 250 patients. Am J Cardiol. 1967 Oct;20(4):457-64. doi: 10.1016/0002-9149(67)90023-9. No abstract available. PMID 6059183
- [Derived] Satilmisoglu MH, Gorgulu S, Aksu HU, Aksu H, Ertas G, Tasbulak O, Buturak A, Kalkan AK, Degirmencioglu A, Koroglu B, Tusun E, Murat A, Oz A. Safety of Early Discharge After Primary Percutaneous Coronary Intervention. Am J Cardiol. 2016 Jun 15;117(12):1911-6. doi: 10.1016/j.amjcard.2016.03.039. Epub 2016 Apr 6. PMID 27156829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process began at May 2013 and finished May 2015. Acibadem University Medical Faculty, Mehmet Akif Ersoy Chest and Cardiovascular Surgery Training and Research Hospital, Dr.Siyami Ersek Chest and Cardiovascular Surgery Training and Research Hospital were the centers involved in the study.Nine-hundred subjects were enrolled.
Pre-assignment Details: 131 patients were excluded due to unsuccesful PPCI, cardiogenic shock, signs of heart failure, stroke within a month, patients treated with thrombolytic agents for the index STEMI,chest pain recurrence, clinically significant arrhythmia >6 hours after PPCI, hypotension (<100 mmHg SBP) persisting after PPCI,inability to get informed consent.
Period: Overall Study
Arm/Group | Early Discharge Group | Standard Discharge Group
Started | 384 | 385
Completed | 370 | 363
Not Completed | 14 | 22
Not completed — Physician Decision | 14 | 22

BASELINE CHARACTERISTICS:
Population: Patients baseline characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Discharge Group | Standard Discharge Group | Total
Number analyzed (Participants) | 370 | 363 | 733
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.55 (10.25) | 54.63 (11.82) | 54.59 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 324 | 316 | 640

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality and Readmission at 30 Days.
Description: The primary end points were all cause mortality by 1 month and readmission due to reinfarction, unstable angina, arrhythmia, congestive heart failure, revascularization, stroke or major bleeding at 1 month.
Time Frame: 30 DAYS
Measure: Number; unit: participants
Arm/Group | Early Discharge Group | Standard Discharge Group
Number analyzed (Participants) | 370 | 363
participants | 16 | 28
Statistical Analysis 1: Comparison: Early Discharge Group vs Standard Discharge Group; Categorical data were analyzed with χ2.Comparisons were also analyzed by χ2 between the early discharge and standard treatment arm for the primary outcomes; Test type: Superiority or Other; p < 0.05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Early Discharge Group: In the early discharge group, patients are actively targeted for hospital discharge within 48-56 hours.
  early discharge: In the early discharge group, patients are actively targeted for hospital discharge within 48-56 hours.
  During 2 year study period, 900 PPCI patients arrived at the three different study centers. 769 patients were randomized in to two groups. There were 384 patients in the early discharge arm. Four patients were excluded due to social repatriation reasons. Furthermore, a total of 10 patients were excluded for follow up reasons such as loosing contact with the patient or refusing to show up in the end of 1 month at the cardiology outpatient clinic. The study was terminated with 370 patients in the early discharge group.
- Standard Discharge Group: Patients who stay longer (96-120 hours) as of a standard procedure. During the two year study period, 900 PPCI patients arrived at the three different study centers. After the exclusion of 131 patients due to primary exclusion criteria 769 patients were randomized in to two groups. There were 385 patients in the standard discharge group. Sixteen patients were excluded due to primary exclusion criteria such as signs of heart failure (n=7, %), clinically significant arrhythmia requiring treatment (n=3, %), chest pain recurrence (n=4,%), cardiogenic shock (n=1,%). Furthermore, a total of 6 patients were excluded for follow up reasons such as loosing contact with the patient or refusing to show up in the end of 1 month at the cardiology outpatient clinic. The study was terminated with 363 patients in the standard discharge group.
Arm/Group | Early Discharge Group | Standard Discharge Group
Serious Adverse Events (participants affected / at risk) | 16/370 | 28/363
Other Adverse Events (participants affected / at risk) | 0/370 | 0/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Discharge Group (N=370) | Standard Discharge Group (N=363)
All cause mortality and readmission (Cardiac disorders) | 16 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No